CLINICAL TRIAL: NCT06168370
Title: Personalized, CT-guided Antithrombotic Therapy Versus Lifelong Single Antiplatelet Therapy to Reduce Thromboembolic and Bleeding Events in Non-atrial Fibrillation Patients After Transcatheter Aortic Valve Implantation: a Pragmatic, International, Multicentre, Randomized Clinical Trial
Brief Title: Personalized, CT-guided Antithrombotic Therapy Versus Lifelong Single Antiplatelet Therapy to Reduce Thromboembolic and Bleeding Events in Non-atrial Fibrillation Patients After Transcatheter Aortic Valve Implantation
Acronym: POP ATLANTIS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Antonius Hospital (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); Pitié-Salpêtrière Hospital (Other)
Responsible Party: Principal Investigator, Jurriën M. ten Berg, MD, PhD, Clinical Professor, St. Antonius Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-504637-42-01
Record Dates: First submitted 2023-10-20; First posted 2023-12-13 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Severe Aortic Valve Stenosis
Keywords: aortic stenosis; bleeding; tavi; ct; personalized antithrombotic therapy; tavr
MeSH Terms: conditions — Aortic Valve Stenosis; Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CT guided strategy (Experimental): The intervention group will undergo CT scan after 3 months. If subclinical valve thrombosis is detected, anticoagulation will be started. If no subclinical valve thrombosis is detected, the SAPT is stopped, unless another indication is present.
  Interventions: Radiation: CT guided strategy
- Standard care (No Intervention): Standard of care with lifelong SAPT after TAVI

INTERVENTIONS:
Radiation: CT guided strategy — 1. With signs of subclinical valve thrombosis on 4D-CT at 3 months after TAVI are switched from SAPT to apixaban. Patients fulfilling the dose reduction criteria according to the drug label, or with a Clinical Frailty Scale ≥4 will receive 2.5mg bid, patients not meeting these criteria will receive a standard dose of 5mg bid.
  2. Without signs of subclinical valve thrombosis on 4D-CT at 3 months after TAVI, without another indication for antiplatelet therapy stop their SAPT.
  3. Without signs of subclinical valve thrombosis on 4D-CT at 3 months after TAVI with another indication for antiplatelet therapy continue life-long SAPT.
  Arms: CT guided strategy

SUMMARY:
The POPular ATLANTIS trial aims to investigate CT-guided antithrombotic therapy compared to lifelong single antiplatelet therapy after a transcatheter aortic valve implantation (TAVI) procedure. Only patients without an indication for anticoagulants will be included in this trial. Currently, lifelong single antiplatelet therapy (mostly aspirin) is considered the standard of care for these patients. However, this approach poses a bleeding risk with only a minimal reduction in thromboembolic events.

After 3 months, a CT scan will be conducted to assess the presence of thrombosis on the newly implanted TAVI valve. Based on the results of a 4D CT scan, the decision will be made whether the patient should receive no anticoagulant or antithrombotic therapy with apixaban. CT-guided antithrombotic therapy holds the potential for a greater reduction in thromboembolic events without increasing the bleeding risk.

ELIGIBILITY:
Inclusion Criteria:

* Successful TAVI (according to the VARC-3 criteria)10 with any approved device
* Ability to understand and to comply with the study protocol
* Written informed consent

Exclusion Criteria:

* Existing indication for oral anticoagulation (e.g. atrial fibrillation, obstructive valve thrombosis detected by echocardiography prior to inclusion)
* Existing indication for dual antiplatelet therapy at three months after TAVI (rare at this time point)
* Creatinine clearance <15 mL/min (based on the CKD-EPI formula) or on renal replacement therapy

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2500 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Thromboembolic events | Through study completion, a median of 2.5 years
  Composite of cardiovascular death, ischaemic stroke, transient ischaemic attack, myocardial infarction, systemic embolism and clinically significant valve thrombosis according to the VARC-3 criteria
All bleeding | Through study completion, a median of 2.5 years
  Defined as the composite of type 1-4 bleeding, according to the VARC-3 criteria

SECONDARY OUTCOMES:
Net clinical benefit, defined as the composite of cardiovascular mortality, stroke, transient ischaemic attack, systemic embolism, clinically significant valve thrombosis and type 1-4 bleeding according to the VARC-3 criteria | Through study completion, a median of 2.5 years
Major bleeding (VARC-3 type 2-4) | Through study completion, a median of 2.5 years
Cerebrovascular events (All stroke and TIA according to VARC-3) | Through study completion, a median of 2.5 years
Cardiovascular mortality | Through study completion, a median of 2.5 years
All-cause mortality | Through study completion, a median of 2.5 years
Aortic bio-prosthetic valve dysfunction assessed by echocardiography yearly after TAVI (standard care), as assessed according the VARC-3 criteria for Bioprosthetic Valve Dysfunction. | Through study completion, a median of 2.5 years
  Bioprosthetic Valve Dysfunction can be split into 'Structural Valve Deterioration' Non-Structural Valve Dysfunction', 'Thrombosis' and 'Endocarditis'. For exact definitions of the sub-groups, VARC-3 criteria can be consulted.
Quality of life as assessed by EuroQol- 5 Dimension 5 Level (EQ-5D-5L) at baseline, 3 and 12 months, and then yearly after TAVI procedure. | Through study completion, a median of 2.5 years
  The EQ-5D-5L is a standardized health-related quality of life instrument that assesses individuals across five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. It generates a health profile that can be converted into a single index value, commonly ranging from -0.594 to 1, where 1 represents full health, 0 indicates a state equivalent to death, and negative values reflect health states perceived as worse than death.
Quality of life as assessed by Kansas City Cardiomyopathy Questionnaire (KCCQ) at baseline, 3 and 12 months, and then yearly after TAVI procedure. | Through study completion, an median of 2.5 years
  The Kansas City Cardiomyopathy Questionnaire (KCCQ) is a disease-specific instrument assessing heart failure patients across domains such as Total Symptoms, Physical Limitation, and Quality of Life, with scores ranging from 0 to 100. Higher scores indicate better health-related quality of life, while lower scores suggest increased symptomatology and functional limitations in heart failure patients.
Quality of life as assessed by Short Form Health Survey (SF-12) at baseline, 3 and 12 months, and then yearly after TAVI procedure. | Through study completion, a median of 2.5 years
  The Short Form 12 (SF-12) is a widely used health survey that measures health-related quality of life across physical and mental domains. It generates two summary scores, the Physical Component Summary (PCS) and the Mental Component Summary (MCS), both ranging from 0 to 100, where higher scores indicate better health status, and these summaries provide a concise assessment of an individual's overall physical and mental well-being.
Medication adherence as assessed by the Medication Adherence Report Scale (MARS-5) yearly after randomization. | Through study completion, a median of 2.5 years
  The Medication Adherence Report Scale (MARS) is a self-report questionnaire designed to assess medication adherence in patients. It consists of five items, and scores range from 1 to 5 for each item, with higher scores indicating better medication adherence. Interpretation involves understanding that higher total scores on the MARS reflect a higher level of adherence to prescribed medications.
Cost-effectiveness assassment of a CT-guided antithrombotic strategy after TAVI using EQ-5D-5L | Through study completion, a median of 2.5 years
  The EQ-5D-5L questionnaire measures health status across five dimensions, providing a standardized index value that is widely used in cost-effectiveness analyses, particularly for estimating Quality-Adjusted Life Years (QALYs) and assessing the impact of healthcare interventions on health-related quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- St. Antonius Hospital, Nieuwegein, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided